CLINICAL TRIAL: NCT03869671
Title: Optimizing Bio-behavioral HIV Prevention Approaches for People Who Inject Drugs
Brief Title: Pre-exposure Prophylaxis (PrEP) for People Who Inject Drugs (PWID)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study design was changed and this clinical trial will not be conducted.
Sponsor: Boston University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-34960; K01DA043412-01A1 (NIH)
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Intravenous Drug Abuse
Keywords: Antiretroviral pre-exposure prophylaxis (PrEP); Syringe exchange program (SEP); HIV-related risk behaviors; Adherence intervention; People who inject drugs (PWID)
MeSH Terms: conditions — Substance Abuse, Intravenous; Adherence Interventions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP uptake/adherence intervention (Experimental): A trained interventionist will deliver the manualized, single session PrEP uptake/adherence intervention in private counseling rooms at a community-based setting.
  Interventions: Behavioral: PrEP uptake/adherence intervention
- Harm reduction standard of care (Active Comparator): Participants will be provided harm reduction supplies and health information and counseling according to routine practice at the community-based setting.
  Interventions: Behavioral: Harm reduction standard of care

INTERVENTIONS:
Behavioral: PrEP uptake/adherence intervention — The interventionist will follow the manual to deliver informational and motivational strategies to participants to enhance their PrEP uptake (including completing clinical screening and obtaining/filling a PrEP prescription) and adherence (taking daily oral PrEP doses). The interventionist will assist participants in problem-solving around topics including limited transportation options, identifying local pharmacies, storing medications given complex living arrangements, coping with side effects, communicating with providers and pharmacists, and maintaining daily medication schedules with reminders and cues.
  Arms: PrEP uptake/adherence intervention
Behavioral: Harm reduction standard of care — Participants will be provided with harm reduction supplies and health information and counseling according to routine practice at the community-based setting (harm reduction organization).
  Arms: Harm reduction standard of care

SUMMARY:
People who inject drugs (PWID) experience high risk of HIV acquisition. Antiretroviral pre-exposure prophylaxis (PrEP) is an efficacious biomedical HIV prevention strategy for high risk HIV-uninfected individuals including PWID, yet uptake has been low in this population and uptake and adherence interventions have not been developed or tested. Drawing from formative qualitative research, the overall goal of this project is to develop an intervention to promote PrEP uptake and adherence among PWID in the U.S. Northeast. The investigators will:

* Analyze existing literature and data to identify specific barriers and facilitators to PrEP uptake and adherence among PWID to inform the initial adaptation of existing theory-based interventions;
* Conduct qualitative interviews with ~30 PWID and ~10 key informants (PrEP and other clinical and social service providers) to identify intervention targets;
* Develop and iteratively refine and finalize an intervention manual based on feedback from qualitative exit-interviews with an interventionist and ~10 PWID; and
* Conduct a pilot randomized clinical trial (RCT) in ~50 HIV-uninfected PWID to compare PrEP uptake and adherence outcomes and assess intervention feasibility and acceptability.

DETAILED DESCRIPTION:
This mixed methods phased research will use qualitative and quantitative techniques to improve PrEP uptake and adherence among PWID through the following three phases:

* Phase 1 will identify the modifiable determinants of PrEP uptake and adherence among HIV-uninfected PWID using in-depth qualitative interviews with PWID and key informants (KIs). Qualitative interviews will explore perceived acceptability and identify barriers and facilitators to PrEP uptake and adherence among ~30 HIV-uninfected PWID and explore perspectives on optimal PrEP delivery methods with ~15 KIs (e.g., PrEP physicians, community-based organization staff members with experience working with PWID).
* Phase 2 will involve identifying intervention targets and adapting existing intervention strategies to improve PrEP uptake and adherence among PWID. This will involve reviewing the literature to identify and select components of existing, evidence-based medication adherence interventions to adapt for the unique determinants of PrEP uptake and adherence among PWID. Investigators will then develop and iteratively refine and finalize an intervention manual by conducting an open-pilot of the intervention in a community-based setting. Refinements will be based on feedback from qualitative exit-interviews with the interventionist and ~10 PWID.
* Phase 3 will involve pilot testing the resulting PrEP uptake and adherence intervention in a selected community-based setting to obtain preliminary data on PrEP uptake and adherence outcomes (primary outcomes) and intervention feasibility and acceptability (secondary outcomes). Investigators will use a pilot RCT design with a mixed methods process evaluation in which 50 HIV-uninfected PWID will be randomized to the PrEP intervention or a control condition (SEP standard of care; n=25 per arm). Investigators will assess changes in PrEP outcomes (primary outcomes of uptake and adherence) and key implementation measures (e.g., secondary outcomes of acceptability, feasibility, adoption by the interventionist).

ELIGIBILITY:
For all phases:

Inclusion Criteria:

* An adult PWID
* Self report of any high risk behaviors for HIV (past-month receptive syringe sharing, transactional sex, condomless sex with an HIV-infected or unknown status partner)

Exclusion Criteria:

* Unable or unwilling to provide informed consent

For Phase 3 (the RCT pilot):

Inclusion Criteria:

* Clinically eligible for PrEP (confirmed HIV-uninfected status, adequate renal function [estimated creatinine clearance ≥60 ml/min], and documented hepatitis B virus [HBV] status)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
PrEP uptake by self-report | 1 month
  measured using 1 item in a structured questionnaire
PrEP uptake by self-report | 3 months
  measured using 1 item in a structured questionnaire
PrEP uptake by pharmacy records | 1 month
  measured by accessing pharmacy records
PrEP uptake by pharmacy records | 3 months
  measured by accessing pharmacy records
PrEP adherence by self-report | 1 month
  measured using 1 item in a structured questionnaire to determine the proportion of doses taken as prescribed
PrEP adherence by self-report | 3 months
  measured using 1 item in a structured questionnaire to determine the proportion of doses taken as prescribed
PrEP adherence by dried blood spot | 1 month
  measured via detection of tenofovir and emtricitabine in dried blood spots (DBS)
PrEP adherence by dried blood spot | 3 months
  measured via detection of tenofovir and emtricitabine in dried blood spots (DBS)

SECONDARY OUTCOMES:
Participant satisfaction with intervention content | 1 month
  assessed via qualitative exit interviews exploring satisfaction with the intervention content (including an open-ended question on topics that were helpful and unhelpful)
Participant satisfaction with intervention delivery methods | 1 month
  assessed via qualitative exit interviews exploring satisfaction with the intervention delivery methods (including an open-ended question on how helpful or unhelpful the intervention delivery methods were)
Interventionist satisfaction with training materials | 1 month
  assessed via qualitative exit interviews exploring satisfaction with the training materials for interventionists (including an open-ended question on how helpful or unhelpful the training materials were)
Interventionist satisfaction with intervention manual | 1 month
  assessed via qualitative exit interviews exploring satisfaction with the intervention manual (including an open-ended question on how helpful or unhelpful the intervention manual was)
Interventionist satisfaction with intervention content | 1 month
  assessed via qualitative exit interviews exploring satisfaction with the intervention content (including an open-ended question on topics that were helpful and unhelpful)
Interventionist satisfaction with intervention delivery methods | 1 month
  assessed via qualitative exit interviews exploring satisfaction with the training materials, intervention manual, intervention content, intervention delivery methods (including an open-ended question on how helpful or unhelpful the intervention delivery methods were)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bazzi, PhD, MPH, Principal Investigator — Boston University

IPD SHARING:
Plan to Share IPD: No